CLINICAL TRIAL: NCT00942058
Title: Serum Carbonic Anhydrase 9 (CA9) Level as Biological Marker of the Treatment Response in Metastatic Renal Cell Cancer : a Pilot Study
Brief Title: Serum CA9 Level as Biological Marker of the Treatment Response in Metastatic Renal Cell Cancer
Acronym: CA9CRM
Status: Terminated | Type: Observational
Why Stopped: Difficult for recruiting
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 0808071; 2008-A01125-50 (Other: AFSSAPS)
Record Dates: First submitted 2009-06-17; First posted 2009-07-20 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Metastatic Kidney Cancer; Metastatic Renal Cell Carcinoma
Keywords: biological markers; CA9 protein; metastatic conventional renal cell cancer; kidney cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CA9 level: Serum and urinary CA9 level
  Interventions: Other: Serum and urinary CA9 level

INTERVENTIONS:
Other: Serum and urinary CA9 level — Blood and urinary samples are collected before treatment and at 1, 3, 6, 9 and 12 months.

SUMMARY:
One third of patients with kidney cancer are diagnosed in the metastatic stage, and among patients with a localized form, about 30 to 40% will develop metastases after surgery.

Medical treatment of metastatic renal cancer include immunotherapy with interferon α and/or IL-2, or targeted therapies such as anti-angiogenic (anti-vascular endothelial growth factor (VEGF), anti-tyrosine kinase inhibitors and m-TOR). These treatments sometimes associated (or IL2 + INF or INF AntiVEGF) do allow for objective response in 15 to 30% of cases (net benefit of targeted therapies), but are carriers of potentially significant side effects and are very expensive. The treatment response is considered on imaging exams repetitive, costly and inconsistently reliable. A serum marker of tumor development would be particularly welcome.

CA9 is an oncogene also know as CA IX, carbonic anhydrase 9 or MN/CA9. The gene encoding an oncoprotein called indifferently membrane antigen MN, MN/CA9 isoenzyme, carbonic anhydrase IX CA9, G250/MN/CA9 or protein G250. It was demonstrated that the level of expression of CA9 in tumor tissue can be used as a predictive marker of response to immunotherapy.

In previous studies, the investigators tried to use CA9 to improve the differential diagnosis of kidney tumors using tumor biopsy or fine needle aspiration. More recently, the investigators have developed the ELISA and quantitative reat time polymerase chain reaction (RT-PCR) to study the CA9 protein and CA9 mRNA in the serum of patients with non-metastatic kidney cancer. The investigators have thus shown that CA9 was overexpressed prior to surgery and that this expression disappeared after tumor ablation.

DETAILED DESCRIPTION:
We propose a pilot study of CA9 serum in patients with adenocarcinoma metastatic cell treated by conventional immunotherapy and / or targeted therapy. This pilot study aims to test the CA9 serum marker of response to medical treatment

ELIGIBILITY:
Inclusion Criteria:

* Conventional renal cell cancer with a pathological diagnosis
* Metastatic disease
* Consent form signed
* social security regimen affiliated

Exclusion Criteria:

* Other cancer treated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a metastatic conventional renal cell cancer. All patients must sign a consent form to be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2009-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
serum protein CA9 and mRNA CA9 level under medical treatment | before treatment, at 1, 3, 6, 9 and 12 months

SECONDARY OUTCOMES:
Correlation clinical response (complete response, partial response, stabilization, progression)-evolution serum CA9 level in blood and urine | Before treatment, at 1, 3, 6, 9, and 12 months
The type and duration of clinical response based on the initial rate and the slope of decline | Before treatment, at 1, 3, 6, 9, and 12 months
serum CA9 level basis and during the following treatment groups of the MSKCC prognostic | Before treatment, at 1, 3, 6, 9, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jacques TOSTAIN, MD-PhD, Study Director — CHU de Saint-Etienne; Nicolas MOTTET, MD, Principal Investigator — CHU de Saint-Etienne
Locations (3):
- France (3):
  - Centre Jean Perrin, Clermont-Ferrand
  - CHU de Saint-Etienne, Saint-Etienne
  - Institut Cancérologique de la Loire, Saint-Priest-en-Jarez

REFERENCES:
- [Background] Li G, Feng G, Gentil-Perret A, Genin C, Tostain J. Serum carbonic anhydrase 9 level is associated with postoperative recurrence of conventional renal cell cancer. J Urol. 2008 Aug;180(2):510-3; discussion 513-4. doi: 10.1016/j.juro.2008.04.024. Epub 2008 Jun 11. PMID 18550116